CLINICAL TRIAL: NCT02599753
Title: Investigating the Microstructural and Functional Alterations of Brain in Parkinson's Disease Patients With Neuropsychiatric Disorders by Multimodal Neuroimaging
Brief Title: Investigating the Microstructural and Functional Alterations of Brain in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Hsin Weng, Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-4874A
Record Dates: First submitted 2015-11-01; First posted 2015-11-09 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ for Parkinson's Disease (Experimental): The participants qualify for the study will return to the clinic at a later date and will have catheter(s) placed for i.v. administration of 18F- DTBZ for injection. The participants will receive a single i.v. bolus of 18F- DTBZ, followed by brain PET imaging of 10 minutes duration, approximately 80 minutes post-dose injection. Vital signs will be obtained prior to and immediately after the administration of 18F- DTBZ, and at the completion of the imaging session. Adverse events will be continuously monitored during the imaging session. The participants experience any adverse event will not be discharged until the event has resolved or stabilized.
  Interventions: Drug: 18-FDTBZ

INTERVENTIONS:
Drug: 18-FDTBZ — During this study, participants will receive a single i.v. administration of approximately 370MBq (10 mCi) 18F- DTBZ immediately prior to imaging. The dosage of DTBZ is 10 nmole. The effective dose in human body is about 5.6 mSV.
  The proposed dose for this study is based on the investigators' phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG (Lin 2010).

SUMMARY:
The objective of this protocol is to investigate the microstructural alterations and monoaminergic function in Parkinson's disease patients with impulse control disorders and cognitive impairment by multimodal MRI and 18F-DTBZ PET imaging.

DETAILED DESCRIPTION:
Study duration is expected to be completed in a period of 4 year. This study will compare the microstructural integrity by multimodal MRI imaging and monoaminergic function by18F- DTBZ PET in 35 PD patients without dementia/ICD (PD group), 35 patients with mild cognitive impairment (PD-MCI), 35 PD patients with dementia (PDD group), and 35 patients with impulse control disorders (PD-ICD group).

ELIGIBILITY:
Inclusion Criteria:

1. PD group: 35 subjects with a diagnosis of PD whom must:

   * Male or female patients, age range 20~80.
   * Patients should not have any clinical evidence of cognitive impairment or ICD.
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
2. PD-MCI group: 35 subjects with a diagnosis of PD with mild cognitive impairment whom must:

   * Male or female patients, age range 20~80.
   * Patients should be fulfilled the"Diagnostic Criteria for Mild Cognitive Impairment in Parkinson's Disease: Movement Disorder Society Task Force Guidelines" as PD-MCI. (Litvan, 2012; Appendix II).
   * Patients should not have any clinical evidence of ICD.
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
3. PDD group: 35 subjects with a diagnosis of PD with dementia whom must:

   * Male or female patients, age range 20~80.
   * Patients should be fulfilled the "Movement Disorders Society diagnostic criteria of PDD as "possible" or "probable" PDD (Emre, 2006). (Appendix III)
   * Patients should not have any clinical evidence of ICD. iv.Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
4. PD-ICD group: 35 subjects with a diagnosis of PD with ICD whom must:

   * Male or female patients, age range 20~80.
   * Patients should be fulfilled one of the diagnostic criteria or definition in these ICDs: pathological gambling, hypersexuality, compulsive shopping, compulsive eating, punding, and compulsive medication use (Voon, 2009). (Appendix IV).
   * Patients should not have any clinical evidence of dementia or cognitive impairment.
   * Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
5. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus, multiple infarction and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
6. Any evidence of secondary parkinsonism (multiple infarcts, intoxication, and hydrocephalus, etc) or other neurodegenerative diseases (multiple system atrophy, progressive supranuclear palsy).
7. History of allergy to radioligands that contain 18F isotope.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The difference of specific uptake ratio (SUR) of 18F- DTBZ between each diagnostic group | 4 years
  The SUVRs of 18F-FP-(+)-DTBZ in ipsilateral caudate, anterior putamen, and bilateral nucleus accumbans were significantly lower in PDD group than those of PD group.

SECONDARY OUTCOMES:
The difference of eigenvalues obtained from diffusion tensor imaging (DTI) between each diagnostic group. | 4 years

OTHER OUTCOMES:
The correlation between SURs of 18F-DTBZ and eigenvalues of DTI in each brain regions and the severity of motor or nonmotor symptoms. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memory Hospital, Taoyuan District, Taiwan